CLINICAL TRIAL: NCT04353869
Title: Targeting Glutamine Metabolism to Prevent Diabetic Cardiovascular Complications
Acronym: GLUTADIAB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: GLUTADIAB
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-03

CONDITIONS: Glutamine; Diabetic; Cardiovascular Complications
Keywords: Diabetes; Cardiovascular complications; Glutamine metabolism
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous blood, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Patients with uncomplicated diabetes and low cardiovascular risk
  During a scheduled hospitalization or consultation as part of the follow-up of their diabetes additions of biological samples, which include:
  A unique venous blood sampling of 9 tubes: 4 x 7 mL EDTA (Éthylènediaminetétraacétique) tubes + 3 x 5 mL EDTA tubes + 2 x 4 mL no additive tubes (total: 51 mL) at a single time during the study and collection of 2 monovettes of 1.6 ml urine (total: 3.2 mL).
  Interventions: Biological: Bio collection
- Group 2: Patients with uncomplicated diabetes and high cardiovascular risk
  During a scheduled hospitalization or consultation as part of the follow-up of their diabetes additions of biological samples, which include:
  A unique venous blood sampling of 9 tubes: 4 x 7 mL EDTA tubes + 3 x 5 mL EDTA tubes + 2 x 4 mL no additive tubes (total: 51 mL) at a single time during the study and collection of 2 monovettes of 1.6 ml urine (total: 3.2 mL).
  Interventions: Biological: Bio collection
- Group 3: Patients with complicated diabetes
  During a scheduled hospitalization or consultation as part of the follow-up of their diabetes additions of biological samples, which include:
  A unique venous blood sampling of 9 tubes: 4 x 7 mL EDTA tubes + 3 x 5 mL EDTA tubes + 2 x 4 mL no additive tubes (total: 51 mL) at a single time during the study and collection of 2 monovettes of 1.6 ml urine (total: 3.2 mL).
  Interventions: Biological: Bio collection

INTERVENTIONS:
Biological: Bio collection — venous blood sampling and collection of urine

SUMMARY:
Experimental data suggest that glutamine catabolism in involved in the activation of macrophages by generating TCA(Tricarboxylic acid) intermediates that promote the pro-inflammatory polarization of macrophages. The project investigates the possible link between glutaminolysis, monocytes polarization and diabetes related cardiovascular complications in humans

DETAILED DESCRIPTION:
The aim of the study is to investigate the role of glutamine metabolism in the pro-inflammatory activation of macrophages in diabetes and related cardiovascular complications.

The study focuses on 3 adult patients' population with different diabetic status and level of cardiovascular risk:

* Patients with uncomplicated type 1 or type 2 diabetes and low cardiovascular risk
* Patients with uncomplicated type 1 or type 2 diabetes and high cardiovascular risk
* Patients with complicated type 1 or type 2 diabetes

Participants (n=975) will be recruited at clinical sites, in the diabetes and cardiology departments (APHP, Bichat - Claude-Bernard Hospital and APHP, Lariboisière Hospital), over a 2-year period.

The study will consist in a single visit. During a scheduled hospitalization or consultation as part of the follow-up of their diabetes or as part of the follow-up of their cardiological problems, clinical data will be collected as well as additional blood and urine samples for analyses and biobanking. There will be no other intervention specific to the study.

ELIGIBILITY:
Inclusion criteria General inclusion criteria applying to the five populations are the following:

* Age above 18 years
* BMI between 25 and 40 kg/m²

Inclusion criteria according to study group are listed below.

Group 1: Patients with uncomplicated diabetes and low cardiovascular risk, additional inclusion criteria are:

* 5 or more years of diabetes
* 6% < HbA1c < 10%
* no history of cardiovascular event, diabetic microvascular complications (kidney function normal and albuminuria/creatininuria < 30 mg/g)
* Coronary artery calcium score < 100 (assessment < 12 months)

Group 2: Patients with uncomplicated diabetes and high cardiovascular risk, additional inclusion criteria are:

* 5 or more years of diabetes
* 6% < HbA1c < 10%
* no history of cardiovascular eventand diabetic nephropathy no more than stage 2 (i.e. GFR ≥ 60 ml/min by MDRD or CKD-EPI formula and albuminuria/creatininuria ≤ 30 mg/g)
* Coronary artery calcium score > 400 (assessment < 12 months)

Group 3: Patients with complicated diabetes, additional inclusion criteria are:

* 5 or more years of diabetes
* 6% < HbA1c < 10%
* A history of cardiovascular event (myocardial infarction, stroke, peripheral vascular disease, or angioplasty) at least 3 months ago

Exclusion Criteria:

* Solid organ or bone marrow transplant patient
* Pregnant or breastfeeding woman
* Absence of free and informed consent
* Non-affiliation to a social security regimen or CMU (universal health coverage)
* Subject deprived of freedom, subject under a legal protective measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Type 1 and 2 diabetic patients and non-diabetic subjects with various levels of cardiovascular risk
Sampling Method: Probability Sample
Enrollment: 995 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Compare the plasma concentrations of glutamine in patients with various levels of cardiovascular (CV) risk. | DAY 1
  plasma concentration of glutamine in each subject.

SECONDARY OUTCOMES:
Study glutamine metabolism in patients with various levels of CV risk | DAY 1
  plasma concentration of glutamate in each treatment group
Study glutamine metabolism in patients with various levels of CV risk | DAY1
  plasma concentration of a-ketoglutarate, fumarate, and succinate in each treatment group
Study glutamine metabolism in patients with various levels of CV risk | DAY 1
  monocyte cytoplasmic concentration of a-ketoglutarate, fumarate and succinate in each treatment group
study the inflammatory status in patients with various levels of CV risk | DAY 1
  plasma concentration of VEGF (Vascular endothelial growth factor) in each treatment group
study the inflammatory status in patients with various levels of CV risk | DAY 1
  plasma concentration of the proinflammatory cytokines IL-1, IL-6, IL-8 (interleukin) and TNF-a (Tumor Necrosis Factor alpha)
study the inflammatory status in patients with various levels of CV risk | DAY 1
  blood concentration of circulating PBMCs (peripheral blood mononuclear cell)
study the monocyte activation status in patients with various levels of CV risk | DAY 1
  frequency of monocyte subsets (CD14++CD16+, CD14++CD16++, CD14+CD16++)
characterize the transcriptomic program through modification gene expression and epigenetic changes related to KDM6B (Lysine Demethylase 6B) and TET2 (Ten-eleven-translocation 2) activity in blood monocytes from patients with various levels of CV risk | DAY 1
  Number of transcript for each gene
characterize the transcriptomic program through modification gene expression and epigenetic changes related to KDM6B and TET2 activity in blood monocytes from patients with various levels of CV risk | DAY 1
  Number of methylated gene loci and their proportion of methylation
characterize the transcriptomic program through modification gene expression and epigenetic changes related to KDM6B and TET2 activity in blood monocytes from patients with various levels of CV risk | DAY 1
  Frequency and level of histone H3K27me (Methylation of lysine 27 on histone H3) methylation

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Diabétologie - Hôpital Lariboisière, Paris, France
  - Diabetologie Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Julla JB, Girard D, Diedisheim M, Saulnier PJ, Tran Vuong B, Bleriot C, Carcarino E, De Keizer J, Orliaguet L, Nemazanyy I, Potier C, Khider K, Tonui DC, Ejlalmanesh T, Ballaire R, Mambu Mambueni H, Germain S, Gaborit B, Vidal-Trecan T, Riveline JP, Garchon HJ, Fenaille F, Lemoine S, Carlier A, Castelli F, Potier L, Masson D, Roussel R, Vandiedonck C, Hadjadj S, Alzaid F, Gautier JF, Venteclef N. Blood Monocyte Phenotype Is A Marker of Cardiovascular Risk in Type 2 Diabetes. Circ Res. 2024 Jan 19;134(2):189-202. doi: 10.1161/CIRCRESAHA.123.322757. Epub 2023 Dec 28. PMID 38152893